CLINICAL TRIAL: NCT00363194
Title: An Open-Label, Two-Period, Randomized, Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of Single Doses of Pazopanib in Cancer Patients
Brief Title: A Two-way Crossover Study Of The Effect Of Food On The Pharmacokinetics Of Pazopanib In Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VEG10005
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: Pazopanib GW786034 Advanced cancer Metastatic cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lead-In cohort (Experimental): In Part 1 of Lead-In cohort, subjects will be dosed with a single dose of pazopanib with a high-fat breakfast to establish safety and tolerability.
  Interventions: Drug: Pazopanib (GW786034)

INTERVENTIONS:
Drug: Pazopanib (GW786034) — Pazopanib (GW786034)

SUMMARY:
This is two-part study (Part I/Part II). Part I is designed to determine the effect of a low and high fat meal on the pharmacokinetics of single dose pazopanib (GW572016). Part II is designed to allow patients continued access to study drug in a multiple dosing regimen. Patients who are receiving clinical benefit on that regimen will go into the long term rollover study VEG105430 provided they are stable for 8 weeks.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of advanced solid tumors that have progressed following treatment with standard agents. Patients may have either measurable disease by RECIST or may be followed by a tumor marker for assessment of disease.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Adequate bone marrow function: ANC greater than or equal to 1,500 mm cubed; Platelets count greater than or equal to 100,000 mm cubed; Hgb greater than or equal to 9 g per dL
* Adequate renal function as determined by a creatinine clearance greater than 50mL per min calculated by the Cockcroft-Gault Formula; Measured creatinine clearance greater than or equal to 50mL per min by 24-hour urine collection will be acceptable in lieu of a calculated value.
* Urine Creatinine Ratio of less than 1 as assessed in a random or spot urine sample.
* Adequate hepatic function: total bilirubin less than or equal to 1.5 times the upper limit of normal; AST and ALT less than or equal to 2.5 times the upper limit of normal.
* PT, INR, PTT less than or equal to 1.2 times upper limit of normal.
* Male or female at least 18 years of age.
* A woman is eligible to enter and participate in the study if she is of: Non-childbearing potential; Childbearing potential, has a negative serum pregnancy test at screening, and agrees to use adequate contraception per protocol. A man with a female partner of childbearing potential is eligible to enter and participate in the study if he uses a barrier method of contraception or abstinence during the study. If sexually active, patients will continue the recommended contraceptive measures for the duration of the treatment and for 28 days following discontinuation of therapy.
* Predicted life expectancy of at least 12 weeks.
* Written informed consent.
* Able to swallow and retain oral medications.

Exclusion criteria:

* Patients with certain heart problems or history of bleeding within a month.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-09-21 (Actual); Primary Completion 2009-06-19 (Actual); Study Completion 2009-06-19 (Actual)

PRIMARY OUTCOMES:
PK parameters: Cmax, tmax, and AUC | Day 1 and Day 15

SECONDARY OUTCOMES:
Safety and tolerability parameters include evaluation of adverse events (AEs), and changes in clinical laboratory, and vital signs assessments under fed and fasted conditions | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Detroit, Michigan

REFERENCES:
- [Background] Heath EI, Chiorean EG, Sweeney CJ, Hodge JP, Lager JJ, Forman K, Malburg L, Arumugham T, Dar MM, Suttle AB, Gainer SD, LoRusso P. A phase I study of the pharmacokinetic and safety profiles of oral pazopanib with a high-fat or low-fat meal in patients with advanced solid tumors. Clin Pharmacol Ther. 2010 Dec;88(6):818-23. doi: 10.1038/clpt.2010.199. Epub 2010 Oct 27. PMID 20980999
- [Background] Heath EI, Forman K, Malburg L, Gainer S, Suttle AB, Adams L, Ball H, LoRusso P. A phase I pharmacokinetic and safety evaluation of oral pazopanib dosing administered as crushed tablet or oral suspension in patients with advanced solid tumors. Invest New Drugs. 2012 Aug;30(4):1566-74. doi: 10.1007/s10637-011-9725-2. Epub 2011 Aug 3. PMID 21811833
- See also: Results for study VEG10005 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/VEG10005?search=study&search_terms=VEG10005#rs